CLINICAL TRIAL: NCT06327217
Title: Long Term Results After Hip Arthroscopy
Status: Not yet recruiting | Type: Observational
Sponsor: Reinier Haga Orthopedisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: OC-2023-009
Record Dates: First submitted 2024-03-06; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Femoro Acetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hip arthroscopy 5-10jr
  Interventions: Radiation: Bilateral hip x-ray; Other: Questionnaires

INTERVENTIONS:
Radiation: Bilateral hip x-ray — Patients will be asked to visit the clinic for a bilateral hip x-ray, in order to evaluate the degree os osteoarthritis.
Other: Questionnaires — Patients will be asked to complete questionnaires on function, quality of life and pain (the modified Harris Hip Score (mHHS), Hip Outcome Score (HOS), the World Health Organisation Quality of Life Questionnaire (WHOWOL) and Visual Analogue Scale (VAS) for pain). One question will be asked: 'How satisfied are you with the results of the surgery?' on a 10-point scale.

SUMMARY:
A common cause of hip joint pain in the young and active population is femoroacetabular impingement (FAI) syndrome. if FAI is left untreated, the changed morphology will have a negative effect on the existing joint and will contribute to the development of osteoarthritis (OA). Hip arthroscopy is the first choice of operative treatment for FAI. While hip arthroscopy improves the patient reported outcome measures (PROMs), the influence of this treatment on the contribution to the development of osteoarthritis after FAI is to the best of our knowledge still unknown.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet all of the following criteria:

Inclusion Criteria:

* Patient who participated in the cohort study;
* At least 5 years of follow up;
* Patient is able to understand the meaning of the study and is willing to sign the Informed Consent Form.

A potential subject who meets any of the following criteria will be excluded from participation in this study:

Exclusion Criteria:

* Patient who has had hip arthroscopy of both sides;
* Patient is unable or unwilling to sing informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from a previous hip arthroscopy cohort study, who are between 5 and 10 years of follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 451 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the degree of osteoarthritis 5 to 10 years after a hip arthroscopy in comparison with the non-operative side. | 5 to 10 years after hip arthroscopy
  To evaluate the degree of osteoarthritis, the Kellgren and Lawrence-scale will be used.
  The scale ranges from 0 to 4:
  A score of 0 indicates that there is no evidence of osteoarthritis A score of 4 indicates end-stage OA, marked by severe sclerosis, joint space narrowing (sometimes bone-on-bone contact), and large osteophytes.

SECONDARY OUTCOMES:
To evaluate the change in degree of osteoarthritis at 5 to 10 years after a hip arthroscopy in comparison with preoperative/perioperative. | 5 to 10 years after hip arthroscopy
  To evaluate the degree of osteoarthritis, the Kellgren and Lawrence-scale will be used.
  The scale ranges from 0 to 4:
  A score of 0 indicates that there is no evidence of osteoarthritis A score of 4 indicates end-stage OA, marked by severe sclerosis, joint space narrowing (sometimes bone-on-bone contact), and large osteophytes.
To report incidence of total hip replacement within 5 to 10 years after a hip arthroscopy. | 5 to 10 years after hip arthroscopy
  survival of the hip arthroscopy (defined by the incidence of total hip replacement) will be presented as a percentage of the total study population.
To determine the functional outcome of patients and, to determine what factors contribute to a good functional outcome 5/10 years after hip arthroscopy. | 5 to 10 years after hip arthroscopy
  Functional outcomes measured with patient reported outcome measures (PROMs) at 5 to 10 years after hip arthroscopy.
To determine the inter-rater and intra-rater agreement of the Kellgren and Lawrence OA score. | 5 to 10 years after hip arthroscopy
  The scale ranges from 0 to 4:
  A score of 0 indicates that there is no evidence of osteoarthritis A score of 4 indicates end-stage OA, marked by severe sclerosis, joint space narrowing (sometimes bone-on-bone contact), and large osteophytes.
To determine patient satisfaction 5-10 years after hip arthroscopy. | 5 to 10 years after hip arthroscopy
  One question on satisfaction will be asked: 'How satisfied are you with the results of the surgery?' on a 10-point scale.
  With 0 being not satisfied and 10 being very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Reinier Haga Orthopedic Center, Zoetermeer, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided